CLINICAL TRIAL: NCT00680056
Title: Randomised Cross-over Study to Compare the Effect of Formoterol Plus Tiotropium Versus Formoterol Monotherapy on Breathlessness, Dynamic Hyperinflation and Exercise Tolerance in Moderate-to-severe Stable COPD Patients
Brief Title: Add-on Effects of Tiotropium Over Formoterol in Exercise Tolerance on Chronic Obstructive Pulmonary Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: J Alberto Neder, Federal University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIOFOR
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Results first posted 2009-12-03 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2009-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Chronic Bronchitis; Pulmonary Emphysema
Keywords: Pulmonary Disease, Chronic Obstructive; Tiotropium; Formoterol; Bronchodilator Agents; Exercise Tolerance; Randomized Controlled Trial [Publication Type]; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchitis, Chronic; Pulmonary Emphysema | interventions — Formoterol Fumarate; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Formoterol plus Placebo (Tiotropium)
  Interventions: Drug: Formoterol plus Placebo (Tiotropium)
- 2 (Experimental): Formoterol plus Tiotropium
  Interventions: Drug: Formoterol plus Tiotropium

INTERVENTIONS:
Drug: Formoterol plus Placebo (Tiotropium) — Formoterol 12mcg-capsules (2x/d) + Placebo (Tiotropium) (1x/d). Double-blind medication will be dispensed in HandiHalers and Aerolisers during 2 weeks.
  Arms: 1
Drug: Formoterol plus Tiotropium — Formoterol 12mcg-capsule (2x/dia) + Tiotropium 18mcg-capsule (1x/d). Double-blind medication will be dispensed in HandiHalers and Aerolisers during 2 weeks.
  Arms: 2

SUMMARY:
The primary objective is to comparatively evaluate the isolated effects of a long-acting beta2-adrenergic (formoterol fumarate 12µg b.i.d. via Aeroliser) and combined with a long-acting anti-cholinergic (tiotropium bromide 18µg o.d via Handihaler) on breathlessness, dynamic hyperinflation and exercise tolerance in patients with advanced, but stable, chronic obstructive pulmonary disease. The study hypothesis is that combining long acting bronchodilators with different action mechanisms would promote synergistic effects on clinical outcomes.

DETAILED DESCRIPTION:
This will be a single center, randomized, double-blind study consisting of two 2-week treatment periods separated by a 5-7 days washout phase without long-acting bronchodilators. Eligible patients who complete the one week screening phase will be randomized to one of two treatment sequences: 1) Formoterol --> Formoterol + Tiotropium or 2) Formoterol + Tiotropium --> Formoterol. During the treatment periods, patients will be allowed to use a short-acting beta2-adrenergic+short-acting anticholinergic as rescue medication (salbutamol+ipratropium via MDI)

ELIGIBILITY:
Inclusion Criteria:

* COPD patients aged ≥ 40 years with stable moderate-to-severe airflow obstruction (FEV1 < 70% and FEV1/FVC ≤ 70% of predicted normal value) post-bronchodilator
* presenting with a long history of smoking (> 20 pack-years) and chronic breathlessness (Baseline Dyspnoea Index total score < 9)

Exclusion Criteria:

* significant cardiovascular disease, hospitalization for COPD exacerbation or presence of a respiratory tract infection within 1 month of screening
* current or childhood asthma
* a history of allergic rhinitis or other atopic disease
* inability to interrupt usual bronchodilator medication
* use of oral steroids within a month before screening
* need for long-term oxygen therapy, arterial oxygen saturation < 85% at rest anemia, hypo- and hyperthyroidism, hyperadrenergic state
* uncontrolled insulin dependent diabetes mellitus, malignancy, or any disease or condition which limits exercise performance other than COPD
* change in inhaled corticosteroid or theophylline use within 1 month prior to screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2007-11; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Alberto Neder, MD, phD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Pulmonary Function and Clinical Exercise Physiology Unit (SEFICE), São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Berton DC, Reis M, Siqueira AC, Barroco AC, Takara LS, Bravo DM, Andreoni S, Neder JA. Effects of tiotropium and formoterol on dynamic hyperinflation and exercise endurance in COPD. Respir Med. 2010 Sep;104(9):1288-96. doi: 10.1016/j.rmed.2010.05.017. Epub 2010 Jun 26. PMID 20580216

RESULTS

PARTICIPANT FLOW:
Recruitment Details: University clinic Period: January-August (2008)
Pre-assignment Details: After screening and before first baseline visit, patients discontinued long-acting β2-agonists and inhaled anticholinergic bronchodilators (run in period).
  50 patients recruited; 33 screened. 7 excluded: 4 due to chronic obstructive pulmonary disease (COPD) exacerbation and 3 due to protocol violation.
Groups:
- Formoterol Plus Placebo (Tiotropium) First: Formoterol + Placebo (Tiotropium) in first intervention period and Formoterol + Tiotropium in second intervention period (after washout period).
- Formoterol Plus Tiotropium First: Formoterol + Tiotropium in first intervention period and Formoterol + placebo in second intervention period (after washout period).
Period: First Intervention
Arm/Group | Formoterol Plus Placebo (Tiotropium) First | Formoterol Plus Tiotropium First
Started | 16 | 17
Completed | 15 | 15
Not Completed | 1 | 2
Not completed — Mainly Exacerbation of COPD | 1 | 2
Period: Washout Period of One Week
Arm/Group | Formoterol Plus Placebo (Tiotropium) First | Formoterol Plus Tiotropium First
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Formoterol Plus Placebo (Tiotropium) First | Formoterol Plus Tiotropium First
Started | 15 | 15
Completed | 12 | 14
Not Completed | 3 | 1
Not completed — Protocol Violation | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Formoterol Plus Placebo (Tiotropium) First | Formoterol Plus Tiotropium First | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 10 | 6 | 16.0
  >=65 years | 6 | 11 | 17.0
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (8.2) | 67.2 (6.8) | 64.9 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 7.0
  Male | 11 | 15 | 26.0
Region of Enrollment [Number; unit: participants]
  Brazil | 16 | 17 | 33.0

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Exercise Tolerance From Baseline at 2 Weeks
Description: Percentage change from baseline in time to the limit of tolerance on a high intensity constant-speed treadmill exercise test (with a speed corresponding to 80% of that obtained during incremental test)
Time Frame: Baseline and after 2 weeks with each treatment
Population: The specific period where the patient received a given treatment were analysed together.
Measure: Mean (Standard Error); unit: Percentage change
Groups:
- Formoterol Plus Placebo (Tiotropium) Treatment: Formoterol + Placebo (Tiotropium) in either first intervention period or second intervention period.
- Formoterol Plus Tiotropium Treatment: Formoterol + Tiotropium in either first intervention period or second intervention period.
Arm/Group | Formoterol Plus Placebo (Tiotropium) Treatment | Formoterol Plus Tiotropium Treatment
Number analyzed (Participants) | 26 | 26
Percentage change | 68 (14) | 124 (27)
Statistical Analysis 1: Comparison: Formoterol Plus Placebo (Tiotropium) Treatment vs Formoterol Plus Tiotropium Treatment; It was calculated a total sample size of a 2x2 cross-over design as 24 for a two-sided t-test achieves 85% power to infer that the mean difference is not zero, the actual mean difference is 20, the standard deviation of the differences is 15, and the significance level is 0.05; Test type: Superiority or Other; p = 0.038, t-test, 2 sided; Mean Difference (Net) = 56, Standard Deviation 60 — Mean difference= Formoterol plus Tiotropium minus Formoterol plus Placebo(Tiotropium)

2. Secondary Outcome: Mean Score on the Transitional Dyspnea Index (TDI)
Description: TDI is a multidimensional clinical instrument developed to provide a comprehensive assessment of change in dyspnea after an intervention, considering three components (functional impairment, magnitude of task, and magnitude of effort). It ranges from -9 (major deterioration) to +9 (major improvement).
Time Frame: After 2 week of each treatment
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Formoterol Plus Tiotropium Treatment: Formoterol + Tiotropium in first intervention period and Formoterol + placebo in second intervention period (after washout period).
Arm/Group | Formoterol Plus Placebo (Tiotropium) Treatment | Formoterol Plus Tiotropium Treatment
Number analyzed (Participants) | 26 | 26
score on scale | 2.9 (2.5) | 3.8 (1.8)
Statistical Analysis 1: Comparison: Formoterol Plus Placebo (Tiotropium) Treatment vs Formoterol Plus Tiotropium Treatment; Test type: Superiority or Other; p = 0.054, t-test, 2 sided; Mean Difference (Net) = 0.88, Standard Deviation 2.39 — Mean difference=Arm 2 minus Arm 1

ADVERSE EVENTS:
Description: Serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Formoterol Plus Placebo (Tiotropium) First | Formoterol Plus Tiotropium First
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No